CLINICAL TRIAL: NCT02507960
Title: (GCC 1202): Tumor Bed Dose Delivery Using a Breast Specific Radiosurgery Device. The Gamma Pod : A Clinical Feasibility Study
Brief Title: The Gamma Pod: A Clinical Feasibility Study Device GCC 1202: The Gamma Pod: A Clinical Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Department of Radiation Oncology, Principal Investigator, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00052062
Record Dates: First submitted 2015-07-16; First posted 2015-07-24 (Estimated); Results first posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pilot Study (Other): The patient will undergo a conventional CT simulation in supine position without the breast immobilization cup. The purpose of the CT simulation is-two-fold: 1) the investigators will see if the TB volume can be accurately delineated and if the TB volume is too large for Gamma Pod boost; and 2) the CT images are used for planning the patient's whole breast irradiation. If, after viewing the CT images and the patient is deemed a study candidate and consents, the participants will receive a second CT-sim and the Gamma Pod TB boost treatment on the same day as described below.
  Interventions: Device: The Gamma Pod; Device: CT simulation

INTERVENTIONS:
Device: The Gamma Pod — Immobilization of breast during radiation.
Device: CT simulation — See arm description

SUMMARY:
In this study, investigators plan to deliver a 8 Gy Tumor Bed (TB) boost using the Gamma Pod™ system followed by a conventional (50Gy in 25 fractions) or hypofractionated (40Gy in 15 fractions) course of whole breast radiation. The clinical target volume receiving 8 Gy will be the surgical cavity as defined by the surgical clips and post-surgical changes + 5 mm. The planning target volume (PTV) will add 5 mm to the clinical target volume to account for geometric uncertainties.

DETAILED DESCRIPTION:
The current standard of care in our clinic when delivering a conventional course of whole breast radiation is to deliver between 60 and 66 Gy to the tumor bed when negative margins are achieved, with the initial ~45-50 Gy delivered to the whole breast and the 10-16 Gy TB boost delivered in 5-8 fractions.The current standard of care in our clinic when delivering a hypofractionated course of whole breast radiation is to deliver between 50 and 52 Gy to the tumor bed when negative margins are achieved, with the initial ~40-42.5 Gy delivered to the whole breast in 15 or 16 fractions respectively followed 10 Gy TB boost delivered in 4 or 5 fractions (total 20). The clinical target volume for the TB boost in this study is quite similar to conventional TB boost. The only difference is that the planning target volume margin is smaller in this study (5 mm instead of 10 mm) due to the reduced set up uncertainties with the breast cup immobilization and localization devices. The current institutional standard is covering the TB + 15 mm dosimetric margin. Since the reproducibility is improved by 5 mm with the aid of the breast immobilization cup, the TB + 10 mm dosimetric margin will be used on this study. Using the radiobiological equivalent dose (BED) formula, {BED = n D(1 + D/(α/β))}, the 8 Gy single fraction dose is equivalent to 16 Gy delivered in 8 fractions. Wherein the BED formula, n is the number of fractions, D is the dose per fraction and α/β is estimated to be between 3 and 4. On this study, the investigators will deliver either 40 Gy in fifteen (15) fractions (hypofractionated) or 50Gy in twenty-five (25) fractions (conventional) to the whole breast following a single 8 Gy boost using the Gamma Pod™. The summed dose to the boost region will be radiobiologically equivalent to a total dose of 52 (hypofractionated) or 66 Gy (conventional).

The safety and feasibility of delivering the boost dose to the tumor bed using a single fraction external beam is supported by past clinical trials. Besides the use of electrons and external beam from a linear accelerator, intracavitary balloons and intraoperative x-rays and electron beams have also been used to deliver a Tumor Bed (TB) boost. In the T A R G I T trial, a single dose of 20 Gy is delivered to the TB using the Intrabeam™ device while the dose drops to between 5 and 7 Gy 1 cm into the normal breast. With long term follow up (median follow-up of 60.5 months), the 5- year local recurrence rate was less than 2 %. In the largest intraoperative electron experience, investigators delivered 9 to 10 Gy in a single treatment prior to whole breast radiation using 9 (million electron volts) electrons. Long-term local control rates and cosmesis appear similar to or better than more conventional techniques. In this proposed study, the investigators plan to deliver 8 Gy to the TB rather than 20 Gy with low energy x-rays or 9-10 Gy with electrons before whole breast irradiation, based on 1) there is no benefit of dose escalation over the biological equivalent dose of 16 Gy at 2 Gy per fraction which is equal to 8 Gy in 1 fraction and 2) known increased side effects with higher doses to the tumor bed. The investigators believe that the proposed dose should be similarly tolerated as observed in these trials, since the volume of normal breast irradiated is similar using a lower dose. In addition, this treatment will similarly shorten treatment by 1 to 1½ weeks by replacing the 8 treatments to the TB.

ELIGIBILITY:
Inclusion Criteria:

* The patient must sign consent for study participation.
* The patient must be female and have a diagnosis of an invasive or non-invasive breast cancer that was treated surgically by a partial mastectomy.
* The patient must be deemed an appropriate candidate for breast conserving therapy (i.e. not pregnant, never had radiation to the treated breast, breast size would allow adequate cosmesis after volume loss from partial mastectomy).
* Patients with involved lymph nodes are candidates for the study as long as regional nodal radiation is not required by the treating physician.
* Surgical margins are negative for invasive or non-invasive breast cancer.
* The greatest dimension of the tumor is less than 4cm before surgery.
* The volume of the TB CTV is less than 25% of the whole breast PTV which is a criteria used for partial breast alone trials (NSABP B-39).
* Multifocal disease is allowed if it was removed by a single lumpectomy resection and the patient remained a candidate for breast conservation.
* Age 60 years and older.
* Women of childbearing potential must use an effective contraceptive method such as condom/diaphragm and spermicidal foam, intrauterine device (IUD), or prescription birth control pills.A negative pregnancy test must be obtained prior to study enrollment or waiver signed.
* The surgical cavity is clearly visible on CT images.
* The patient must weigh less than 150Kg (330lb), which is the limit of the imaging couch.
* The patient must feel comfortable in the prone position.

Exclusion Criteria:

* Patients with proven multicentric carcinoma (tumors in different quadrants of the breast or tumor separated by at least 4 cm).
* Prior radiation therapy above the umbilicus
* Unable to fit into the immobilization breast cup with an adequate seal
* Male gender.
* Patient cannot comfortably be set up in the prone position (i.e. physical disability)
* Unable to fit into the breast immobilization device due to breast size or other anatomical reason.
* Mastectomy is the surgery performed.
* Patient has received prior radiotherapy to the involved breast.
* Regional nodal irradiation is part of the treatment plan.
* Tumor bed is less than 5 mm from the skin surface.
* Patients with skin involvement, regardless of tumor size.
* Patients with connective tissue disorders specifically systemic lupus erythematosis, scleroderma, or dermatomyositis.
* Patients with psychiatric or addictive disorders that would preclude obtaining informed consent.
* Patients who are pregnant or lactating due to potential exposure of the fetus to RT and unknown effects of RT to lactating females.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2018-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M Nichols, MD, Principal Investigator — University of Maryland, Baltimore
Locations (4):
- United States (4):
  - Ummc Msgccc, Baltimore, Maryland
  - Upper Chesapeake Health, Bel Air, Maryland
  - Central Maryland Oncology Center, Columbia, Maryland
  - Baltimore Washington Medical Center, Glen Burnie, Maryland

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pilot Study
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pilot Study
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 10
Age, Continuous [Mean (Full Range); unit: years] | 66.8 [60 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity/Race: White | 15
  Ethnicity/Race: African American | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Demonstration of the Feasibility and Safety of Delivering a Radiation Treatment Using the GammaPod (TM)
Description: Patients must be undergoing breast conserving therapy and PI will evaluate for feasibility by ensuring coverage of the target volume with appropriate dose homogeneity and conformity as defined in the study. Per inclusion criteria, the volume of the tumor bed clinical target volume (CTV) is less than 25% of the whole breast planning target volume (PTV) which is a criteria used for partial breast alone trials (ie. NSABP B-39). If the tumor bed cannot fit this criteria, then patient is unable to be treated utilizing GammaPod.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Study
Number analyzed (Participants) | 17
Participants | 14

2. Secondary Outcome: Number of Participants With Acute Toxicities Measured by Common Terminology Criteria for Adverse Events (CTCAE); The Evaluation of Acute Toxicity During and up to 1 Month After Gamma Pod TB Boost.
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Study
Number analyzed (Participants) | 17
Participants | 14

3. Secondary Outcome: Number of Participants With Long-term Toxicities Measured by Common Terminology Criteria for Adverse Events (CTCAE); The Evaluation of Long-term Toxicity at One Year to Assess the Presence of Subcutaneous Fibrosis and Fat Necrosis.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Study
Number analyzed (Participants) | 17
Participants | 0

4. Secondary Outcome: Efficacy of Medical Adhesive; Number of Participants With Adverse Events From the Use of the Adhesive Spray
Description: Adverse events from the use of the adhesive spray was measured by photos taken pre-entry and during radiation.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Study
Number analyzed (Participants) | 17
Participants | 1

ADVERSE EVENTS:
Time Frame: AEs were collected during radiation treatments and during the follow-up time period (per protocol), approximately a duration of 1 year.
Description: Systematic assessment during through regular physician assessments.
Arm/Group | Pilot Study
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 14/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pilot Study (N=17)
Fatigue (General disorders) | 10
Dermatitis (Skin and subcutaneous tissue disorders) | 11
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 3
Breast Pain (Musculoskeletal and connective tissue disorders) | 4
Limb Edema (General disorders) | 1
Nausea (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-07): https://cdn.clinicaltrials.gov/large-docs/60/NCT02507960/Prot_SAP_000.pdf